CLINICAL TRIAL: NCT00565617
Title: A Pilot Safety and Efficacy Study of Epidural Prefrontal Cortical Stimulation (EpCS) in Severe Treatment Resistant Depression
Brief Title: Epidural Cortical Stimulation for Depression
Acronym: EpCS-D
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Medtronic (Industry); National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Principal Investigator, E. Baron Short, Principal Investigator, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR - 16908
Record Dates: First submitted 2007-11-29; First posted 2007-11-30 (Estimated); Results first posted 2017-09-18 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Treatment Resistant Depression
Keywords: depression; epidural; cortical stimulation; brain stimulation; treatment-resistant; deep brain stimulation; TMS; DBS; ECS
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depression

STUDY DESIGN:
Intervention Model Description: We are currently monitoring participants that were implanted with Epidural Cortical Stimulators starting back in 2008. Primary investigation is completed, but they have implanted devices for investigational treatment of depression. We will keep the study open while they are monitored.
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Synergy, Epidural cortical stimulation (Experimental): Epidural cortical stimulation (medial prefrontal cortex) for treatment resistant depression. The primary aim of this pilot study was to assess the feasibility and safety of EpCS in patients with treatment-resistant depression. Ultimately, for EpCS to be found effective, a much larger double blind placebo controlled study would be needed.
  Interventions: Device: Synergy, Epidural cortical stimulation

INTERVENTIONS:
Device: Synergy, Epidural cortical stimulation — Epidural cortical stimulation
  Other Names: Epidural cortical stimulation

SUMMARY:
Objective: Chronic epidural cortical stimulation (ECS) involves the neurosurgical placement of an electric wire on the surface of the brain with intermittent activation. Over time, ECS modulates local and distal connected brain regions. It is being currently applied over the motor cortex to treat intractable pain. Because of the important role played by the medial prefrontal cortex in mood regulation, the goal of this study is to apply this minimally invasive neurostimulation modality over medial prefrontal cortex in severely ill depressed subjects who have failed all other attempts at treatment.

DETAILED DESCRIPTION:
Hypothesis: Severely Treatment Resistant Unipolar Depressed Subjects with EpCS of medial prefrontal cortex will show a significant decrease in depression symptoms at 6 months post-implant when compared to baseline and to a matched control group treated with electroconvulsive therapy (ECT).

Method: We will enroll 5 subjects with severe refractory depression in an open trial with a 1 month placebo lead in, and for up to 1 years. We will also naturalistically follow 5 matched control patients treated with ECT. Depressive and cognitive symptoms will be rated periodically to assess the safety and efficacy of this procedure.

Significance: This study takes advantage of the expertise at MUSC with various neuromodulation technologies to begin answering the crucial role of targeted cortical brain stimulation and its potential role in treatment resistant depression. This is a crucial pilot study that might lead to an entire new class of therapies for depression.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for this study, a subject must meet all the following inclusion and exclusion criteria:

* Subject has a diagnosis of chronic (≥ two years) or recurrent (multiple prior episodes) depression and is currently experiencing a major depressive episode without psychotic features as defined by DSM IV criteria.
* Subjects may have a diagnosis or unipolar or bipolar depressive episode.
* Subject has not had an adequate response to 4 or more adequate antidepressant treatments in the current depressive episode according to the Antidepressant Treatment History Form (ATHF) (Sackeim et al 1997).
* Subject must be between the ages of 21 and 80.
* Baseline HDRS 24-item ≥ 20 (both visits 1 week apart)
* Subject must be able to complete the evaluations needed for this study including the functional imaging scans.
* Subject must have had a history of one successful course of ECT in the past.
* Subject must provide written informed consent.
* Subject is stable on all antidepressant medication for at least 4 weeks before the baseline visit or not be taking antidepressant medication prior to entering the study.
* Subject must be able to remain on current medication schedule for the first 19 weeks of the study.
* Subject is not on a medication known to increase the risk of cortical stimulation-induced seizures. These include theophylline, stimulant medications, bupropion, or supraphysiological doses of thyroid supplements.

Exclusion Criteria:

The presence of any of the following will exclude a subject from the study:

* The EpCS would (in the investigator's judgment) pose an unacceptable surgical or medical risk for the patient (including, but not limited to: history of serious cardiac or pulmonary problems, stroke, significant brain malformation, progressive neurological disease, central nervous system disease or injury, history of seizure, previous neurosurgical procedure with suspected brain tissue scarring that would increase the risks for seizure or cervical fracture).
* Subject received general anesthetic within the last 30 days prior to enrollment (not including ECT procedure).
* Subject currently has another investigational device or cardiac pacemaker, implantable defibrillator, or other implantable stimulator
* Subject on anticoagulant drugs, with low platelets counts or have PT or PTT abnormalities or other risk factors for intra-operative or post-operative bleeding
* Subject is expected to require full body magnetic resonance imaging (MRI) during the clinical study.
* Subject is judged by the investigator to be acutely suicidal (e.g. within the 30 days prior to the EpCS implant, the subject has made a suicide attempt or gesture or has made specific plans or preparation to commit suicide).
* Subject has a history of schizophrenia, schizoaffective disorder, or other psychotic disorder, active substance abuse or dependence (with the exception to caffeine and nicotine abuse) or a current major depressive episode that includes psychotic features (commonly referred to as psychotic depression) according to the DSM IV criteria.
* Subject with a diagnosis of dementia with a Mini-Mental State Exam (MMSE) ≤23.
* Female subjects with a positive urine pregnancy test.
* Subject with a positive urine drug screen or current alcohol or substance abuse other than nicotine and caffeine.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-10; Primary Completion 2009-12 (Actual); Study Completion 2028-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Edward B Short, MD, MSCR, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided
We are currently monitoring participants. Primary investigation is completed, but they have implanted devices for investigational treatment of depression. We will keep the study open while they are monitored.

REFERENCES:
- [Result] Nahas Z, Anderson BS, Borckardt J, Arana AB, George MS, Reeves ST, Takacs I. Bilateral epidural prefrontal cortical stimulation for treatment-resistant depression. Biol Psychiatry. 2010 Jan 15;67(2):101-9. doi: 10.1016/j.biopsych.2009.08.021. PMID 19819427
- [Result] Williams NR, Short EB, Hopkins T, Bentzley BS, Sahlem GL, Pannu J, Schmidt M, Borckardt JJ, Korte JE, George MS, Takacs I, Nahas Z. Five-Year Follow-Up of Bilateral Epidural Prefrontal Cortical Stimulation for Treatment-Resistant Depression. Brain Stimul. 2016 Nov-Dec;9(6):897-904. doi: 10.1016/j.brs.2016.06.054. Epub 2016 Jun 28. PMID 27443912
- See also: Brain Stimulation Service / Mood Disorders Program at MUSC — https://muschealth.org/medical-services/psychiatry/brain-stimulation
- See also: NARSAD — http://www.narsad.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Epidural Cortical Stimulation Device for Depression: Epidural cortical stimulation device (medial prefrontal cortex), implanted with leads bilaterally at Brodmanns area 10 and 46.
  Synergy, Epidural cortical stimulation: Epidural cortical stimulation. Constant voltage device which can apply varying currents, pulsewidths, frequencies, and duty cycles.
Period: Overall Study
Arm/Group | Epidural Cortical Stimulation Device for Depression
Started | 6
Completed | 5
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Epidural Cortical Stimulation for Depression: Epidural cortical stimulation device (medial prefrontal cortex), implanted with leads bilaterally at Brodmanns area 10 and 46.
  Synergy, Epidural cortical stimulation: Epidural cortical stimulation. Constant voltage device which can apply varying currents, pulsewidths, frequencies, and duty cycles.
  For further description of arm please refer to published paper Ziad Nahas, Berry S. Anderson, Jeff Borckardt, Ashley B. Arana, Mark S. George, Scott T. Reeves, and Istvan Takacs "Bilateral Epidural Prefrontal Cortical Stimulation for Treatment- Resistant Depression" Biological Psychiatry. 2010
Arm/Group | Epidural Cortical Stimulation for Depression
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: HDRS-24 Items
Description: Hamilton Depression Rating Scale (HDRS) is a standard, validated depression rating scale.
  It is a 24 item scale, but the primary score is based on the first 17 answers for a total score for depression.
  0-7=Normal 8 - 13 = Mild Depression 14-18 = Moderate Depression 19 - 22 = Severe Depression > 23 = Very Severe Depression
Time Frame: 7 months from baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Epidural Cortical Stimulation for Depression: Epidural cortical stimulation device (medial prefrontal cortex), implanted with leads bilaterally at Brodmanns area 10 and 46.
  Synergy, Epidural cortical stimulation: Epidural cortical stimulation. Constant voltage device which can apply varying currents, pulsewidths, frequencies, and duty cycles.
Arm/Group | Epidural Cortical Stimulation for Depression
Number analyzed (Participants) | 5
units on a scale
  Pre | 28.4 (8)
  7 months | 13 (11.4)
Statistical Analysis 1: Comparison: Epidural Cortical Stimulation for Depression; Test type: Superiority or Other; p = 0.009, ANOVA

ADVERSE EVENTS:
Arm/Group | Epidural Cortical Stimulation for Depression
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 5/5
Other Adverse Events (participants affected / at risk) | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Epidural Cortical Stimulation for Depression (N=5)
Infection (Infections and infestations) | 1
Hospitalizations (Psychiatric disorders) | 5 — All 5 participants did have hospitalizations for periods of worsening depression and suicidality or inability to care for self. They were all successfully stabilized inpatient and subsequently discharged. This was reported to the FDA. All stable now.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No